CLINICAL TRIAL: NCT00097253
Title: Psychoneuroimmunology and Mind-Body Medicine: Olfaction, Mood, and Physiological Responses
Brief Title: The Effects of Smell on Mood and Physical Responses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Janice K. Kiecolt-Glaser, PhD, The Ohio State University, Department of Psychiatry
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT002122-01 (NIH)
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Stress; Anxiety; Depression
Keywords: Aromatherapy; Smell
MeSH Terms: conditions — Anxiety Disorders; Depression; Anosmia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lavender (Experimental)
  Interventions: Behavioral: Exposure to relaxant and stimulant odors
- Citrus (Experimental)
  Interventions: Behavioral: Exposure to relaxant and stimulant odors
- Water (Placebo Comparator)
  Interventions: Behavioral: Exposure to relaxant and stimulant odors

INTERVENTIONS:
Behavioral: Exposure to relaxant and stimulant odors — A yellow-tinted cotton ball containing 100 ml of the essential oil or distilled water was taped between the nose and upper lip on top of a piece of surgical tape; use of the barrier tape avoided percutaneous absorption . This method provided continuous and uniform exposure across subjects that would not have been possible with ambient room inhalation, and helped maintain experimenter blindness.
  Other Names: Citrus: lemon.

SUMMARY:
The purpose of this study is to examine the body's response to relaxing and stimulating fragrances commonly used in aromatherapy.

DETAILED DESCRIPTION:
Despite aromatherapy's popularity, efficacy data are scant, and potential mechanisms are controversial. This randomized controlled trial examined the psychological, autonomic, endocrine, and immune consequences of one purported relaxant odor (lavender), one stimulant odor (lemon), and a no-odor control (water), before and after a stressor (cold pressor); 56 healthy men and women were exposed to each of the odors during three separate visits. To assess the effects of expectancies, participants randomized to the "blind" condition were given no information about the odors they would smell; "primed" individuals were told what odors they would smell during the session, and what changes to expect. Experimenters were blind.

In each case we measured several different aspects of the cellular immune response, as well as skin barrier repair following tape stripping. This design allowed us to examine the ability of the odors to modulate endocrine and immune function, and health-relevant cutaneous responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with a normal sense of smell

Exclusion Criteria:

* Treatment with medication that has immunological or endocrinological consequences
* Chronic health problems that affect immune or endocrine systems
* Allergy to perfume or cosmetics
* Problems with sense of smell
* Respiratory problems
* Smoker
* Current active asthma
* Use of psychoactive drugs or mood-altering medication
* History of anxiety disorder, major depression, bipolar disorder, schizophrenia, or other psychotic disorders
* History of chest pain or ventricular fibrillation

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2005-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Kiecolt-Glaser, PhD, Principal Investigator — Ohio State University Institute for Biobehavioral Medicine Research
Locations (1):
- Ohio State University Institute for Biobehavioral Medicine Research, Columbus, Ohio, United States

REFERENCES:
- [Result] Kiecolt-Glaser JK, Graham JE, Malarkey WB, Porter K, Lemeshow S, Glaser R. Olfactory influences on mood and autonomic, endocrine, and immune function. Psychoneuroendocrinology. 2008 Apr;33(3):328-39. doi: 10.1016/j.psyneuen.2007.11.015. PMID 18178322
- See also: Related Info — http://www.stressandhealth.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through ads posted in the Columbus, Ohio area.
Pre-assignment Details: We excluded individuals taking cardiovascular medications or medications with obvious immunological or endocrinological consequences. Additional exclusion criteria included perfume allergies, smoking, problems with smell/taste, respiratory problems, asthma, excessive alcohol/caffeine use.
Groups:
- Lavender Oil / Lemon Oil / Water Control: A yellow-tinted cotton ball containing 100 μL of the essential oil or water placebo was taped between the nose and upper lip. Within-subject design was used; each subject was exposed to each of the three odors (lemon, lavender, no odor).
Period: Lavender
Arm/Group | Lavender Oil / Lemon Oil / Water Control
Started | 56
Completed | 56
Not Completed | 0
Period: Lemon
Arm/Group | Lavender Oil / Lemon Oil / Water Control
Started | 56
Completed | 56
Not Completed | 0
Period: Water (Control)
Arm/Group | Lavender Oil / Lemon Oil / Water Control
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lavender Oil / Lemon Oil / Water Control
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.41 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Cortisol and Catecholamine Production
Description: Cortisol, norepinephrine, epinephrine measured before and after physical (cold pressor) stressor, which occurred at 11:00.
Time Frame: 3 Visits with at least 2 weeks between each. Average time to complete all visits was 64.46 days (SD 48.4). Cortisol: 9:05, 10:05, 10:55, 11:45, 12:15, 13:00. Nor/Epi: 9:05, 10:05, 10:55, 11:05, 11:45, 12:15
Measure: Mean (Standard Deviation); unit: pg/ml (log 10)
Groups:
- Lavender: A yellow-tinted cotton ball containing 100 μL of the essential oil or water placebo was taped between the nose and upper lip. Within-subject design was used; each subject was exposed to each of the three odors (lemon, lavender, no odor).
- Water Control; Lemon: A yellow-tinted cotton ball containing 100 μL of water was taped between the nose and upper lip. Within-subject design was used; each subject was exposed to each of the three odors (lemon, lavender, no odor).
Arm/Group | Lavender | Water Control | Lemon
Number analyzed (Participants) | 56 | 56 | 56
pg/ml (log 10)
  Cortisol (post stress) | 0.107 (0.056) | 0.119 (0.071) | 0.107 (0.056)
  Epinephrine (post stress) | 43.5 (32.7) | 44.3 (24.2) | 38.3 (17.9)
  Norepinephrine (Change pre to post stress) | 0.03 (0.02) | 0.03 (0.01) | 0.073 (0.024)
Statistical Analysis 1: Comparison: Lavender vs Water Control vs Lemon; Cortisol. Analyses consisted of repeated-measures linear models fit to each dependent variable.IVs assessed in each model were odor, time, gender, expectancy group (primed vs. blind), their interactions;baseline level of the DV was included as a covariate. Post hoc tests were used as appropriate. A two-sided significance level of alpha = 0.05 was used. Model controlled for Time 1 baseline; Test type: Superiority or Other; p = 0.83, Regression, Linear
Statistical Analysis 2: Comparison: Lavender vs Water Control vs Lemon; Epinephrine. Analyses consisted of repeated-measures linear models fit to each dependent variable.IVs assessed in each model were odor, time, gender, expectancy group (primed vs. blind), their interactions;baseline level of the DV was included as a covariate. Post hoc tests were used as appropriate. A two-sided significance level of alpha = 0.05 was used. Model controlled for Time 1 baseline; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis
Statistical Analysis 3: Comparison: Lavender vs Water Control vs Lemon; Norepinephrine. Model controlled for Time 1 baseline. Comparing timepoints 4 and 5 for pre versus post stressor, e.g. lemon versus water control; Citrus(5-4)-Water(5-4); Test type: Superiority or Other; p = 0.017, Mixed Models Analysis

2. Primary Outcome: Immune Function
Description: Stimulated Cytokine Production (Interleukin-6 (IL-6), Interleukin-10 (IL-10)) measured before and after cold pressor stressor, which occurred at 11:00.
Time Frame: 3 Visits with at least 2 weeks between each. Average time to complete all visits was 64.46 days (SD 48.4). 9:05, 10:05, 11:45
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lavender | Water Control | Lemon
Number analyzed (Participants) | 56 | 56 | 56
pg/ml
  IL-6 | 3.706 (0.814) | 3.622 (0.857) | 3.623 (0.904)
  IL-10 | 1.777 (0.480) | 1.734 (0.463) | 1.787 (0.458)
Statistical Analysis 1: Comparison: Lavender vs Water Control vs Lemon; IL-6. Mixed effect linear models were used to test the hypothesis. These models included the post-odor and post-stress dependent variable measurements with a covariate for the baseline pre-odor measurement. Base 10 logarithms were used for each dependent variable and baseline covariate; Test type: Superiority or Other; p = 0.10, Mixed Models Analysis
Statistical Analysis 2: Comparison: Lavender vs Water Control vs Lemon; IL-10. Mixed effect linear models were used to test the hypothesis. These models included the post-odor and post-stress dependent variable measurements with a covariate for the baseline pre-odor measurement. Base 10 logarithms were used for each dependent variable and baseline covariate; Test type: Superiority or Other; p = 0.50, Mixed Models Analysis

3. Primary Outcome: Skin Barrier Repair
Description: TEWL (Transepidermal Water Loss, via tape stripping procedure)measured before and after cold pressor stressor (11:00). After obtaining baseline measurements on volar forearm, cellophane tape(3M Scotch-type; St. Paul, MN) was applied repeatedly (6-50 times) to remove superficial layer of cornified skin cells. Tape stripping stopped when TEWL was elevated from the basal level of 5-7 g/h/m2 to at least 20 g/h/m2. The number of strips required to reach TEWL X20 g/m2/h was the measure of barrier. TEWL was measured with a computerized evaporimetry instrument, the DermaLabs (CyberDERM, Media, PA).
Time Frame: 3 Visits with at least 2 weeks between each. Average time to complete all visits was 64.46 days (SD 48.4).10:05, 11:45, 13:15
Measure: Mean (Standard Deviation); unit: number tape strips
Groups:
- Lavender; Lemon: A yellow-tinted cotton ball containing 100 μL of the essential oil or water control was taped between the nose and upper lip. Within-subject design was used; each subject was exposed to each of the three odors (lemon, lavender, no odor).
Arm/Group | Lavender | Water Control | Lemon
Number analyzed (Participants) | 56 | 56 | 56
number tape strips
  Time 1 Pre-Stress | 23.21 (11.52) | 24.33 (10.61) | 22.11 (10.47)
  Time 2 Post-Stress | 15.64 (4.76) | 17.78 (7.30) | 16.82 (6.10)
Statistical Analysis 1: Comparison: Lavender vs Water Control vs Lemon; Repeated-measures mixed effects models were used. Model was fit to the log-transformed data. Analysis applied to odor category, e.g. lavender / lemon / water; Test type: Superiority or Other; p = 0.60, Mixed Models Analysis

4. Primary Outcome: Immune Function: Delayed Hypersensitivity to Candida(DTH)
Description: DTH memory responses to a common infectious agent provided a measure of T-cell immunity. Nurses inoculated subject's arm with 0.1ml Candida (stock solution diluted 1:20 in saline, Greer Labs, NC) intradermally, after the cold pressor stressor. The wheal diameter (2 dimensions) was self-assessed at 24, 48, and 72 hours by participants given detailed instructions and templates for measurement.
Time Frame: Day 1 11:45, Day 2 (24h) 11:45, Day 3 (48h) 11:45, Day 4 (72h) 11:45.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Lavender | Water Control | Lemon
Number analyzed (Participants) | 56 | 56 | 56
mm^2 | 10.84 (10.01) | 17.39 (15.08) | 12.40 (10.12)
Statistical Analysis 1: Comparison: Lavender vs Water Control vs Lemon; The maximum DTH wheal of days 1-3 (24, 48, or 72 h) was used as the dependent variable for each subject at each visit. Visits for subjects with a maximum DTH wheal of 5mm or less were excluded. A repeated measures linear model was used to evaluate odor and placebo effects; Test type: Superiority or Other; p = 0.014, Regression, Linear

ADVERSE EVENTS:
Description: No serious or other adverse events were observed.
Arm/Group | Lavender Oil / Lemon Oil / Water Control
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No